CLINICAL TRIAL: NCT05996874
Title: Investigation of the Effect of Dosing Conditions on the Pharmacokinetics of New Oral Semaglutide Formulation in Healthy Participants
Brief Title: A Research Study Comparing the Effect of Different Dosing Conditions on Blood Levels of Semaglutide in a New Tablet Composition in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9924-4977; U1111-1281-4819 (Other: World Health Organization (WHO)); 2022-002848-52 (EudraCT Number)
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Healthy Participants
MeSH Terms: interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Semaglutide: 50 mL water and 30 minutes post-dose fasting (Experimental): Participants will receive oral semaglutide D once daily for 10 days. Dose 1 of oral semaglutide D will be administered for the first 5 days followed by Dose 2 of oral semaglutide D for another 5 days with 50 mL water and 30 minutes post-dose fasting.
  Interventions: Drug: Semaglutide
- Semaglutide: 120 mL water and 30 minutes post-dose fasting (Experimental): Participants will receive oral semaglutide D once daily for 10 days. Dose 1 of oral semaglutide D will be administered for the first 5 days followed by dose 2 of oral semaglutide D for another 5 days with 120 mL water and 30 minutes post-dose fasting.
  Interventions: Drug: Semaglutide
- Semaglutide: 50 mL water and 60 minutes post-dose fasting (Experimental): Participants will receive oral semaglutide D once daily for 10 days. Dose 1 of oral semaglutide D will be administered for the first 5 days followed by Dose 2 of oral semaglutide D for another 5 days with 50 mL water and 60 minutes post-dose fasting.
  Interventions: Drug: Semaglutide
- Semaglutide: 120 mL water and 60 minutes post-dose fasting (Experimental): Participants will receive oral semaglutide D once daily for 10 days. Dose 1 of oral semaglutide D will be administered for the first 5 days followed by Dose 2 of oral semaglutide D for another 5 days with 120 mL water and 60 minutes post-dose fasting.
  Interventions: Drug: Semaglutide
- Semaglutide: 50 mL water and 120 minutes post-dose fasting (Experimental): Participants will receive oral semaglutide D once daily for 10 days. Dose 1 of oral semaglutide D will be administered for the first 5 days followed by Dose 2 of oral semaglutide D for another 5 days with 50 mL water and 120 minutes post-dose fasting.
  Interventions: Drug: Semaglutide
- Semaglutide: 120 mL water and 120 minutes post-dose fasting (Experimental): Participants will receive oral semaglutide D once daily for 10 days. Dose 1 of oral semaglutide D will be administered for the first 5 days followed by Dose 2 of oral semaglutide D for another 5 days with 120 mL water and 120 minutes post-dose fasting.
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Semaglutide — Participants will receive Dose 1 oral semaglutide D for the first 5 days followed by Dose 2 of oral semaglutide D for another 5 days.

SUMMARY:
In this study, a known medicine called 'semaglutide' will be tested in a new tablet version. The medicine will be tested in healthy men to explore the effect of different water volumes and tablet-meal delays on blood levels of semaglutide after 10 days of oral administration. Semaglutide tablets, under the brand name Rybelsus, are approved in the EU and USA for the treatment of type 2 diabetes. Participants will get a daily treatment with dose 1 new oral semaglutide tablet for 5 days followed by another 5 days with a daily treatment of dose 2 new oral semaglutide tablet. Participants will get one tablet each day for 10 days. The tablet should be taken in the morning on an empty stomach with either 50 milliliter (mL) or 120mL water, after an overnight fast of at least 6 hours (no food or drinks). Water is not allowed from 2 hours before dosing. A predefined breakfast will be served either 30, 60 or 120 minutes after taking tablet, depending on the treatment received. Breakfast will need to be eaten within 30 minutes. Which treatment participants will get is decided by chance. The study will last for about 11 weeks. This will include a screening period (up to 28 days), a treatment period (10 days) and a follow-up visit (at least 5 weeks after the last dose). Participants should not take any prescription or non-prescription medicines or herbal products (including St John's wort) within 14 days prior to the screening visit and until the follow-up visit, except for routine vitamins, medicines applied on the skin and occasional use of paracetamol (a mild pain killer). No oral medication can be taken from 2 hours before and, depending on the group participants are in, until 30, 60 or 120 minutes after each dosing with semaglutide.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.5 and 29.9 kilograms per meter square (kg/m^2) (both inclusive)
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator

Exclusion Criteria:

* Glycated Hemoglobin (HbA1c) greater than or equal to (>=) 6.5 percent (%) (48 millimoles per mole [mmol/mol]) at screening
* Use of tobacco and nicotine products, defined as any of the below:

  1. Smoking more than 5 cigarettes or the equivalent per day
  2. Not willing to refrain from smoking and use of nicotine substitute products within 48 hours prior to and during the inpatient periods
* Presence of clinically significant gastrointestinal disorders potentially affecting absorption of drugs and/or nutrients, as judged by the investigator
* Personal or first-degree relative(s) history of multiple endocrine neoplasia type 2 or medullary thyroid carcinoma
* History of major surgical procedures involving the stomach potentially affecting absorption of trial products (e.g. subtotal and total gastrectomy, sleeve gastrectomy, gastric bypass surgery) or current presence of gastrointestinal implant

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2023-08-12 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2024-04-18 (Actual)

PRIMARY OUTCOMES:
AUC0-24h,sema,Day10: Area under the semaglutide plasma concentration-time curve during a dosing interval after the 10th dosing | From 0 to 24 hours after dosing on day 10
  Measured in hour*nanomoles per liter (h*nmol/L).

SECONDARY OUTCOMES:
Cmax,0-24h,sema,Day10: Maximum semaglutide plasma concentration after the 10th dosing | From 0 to 24 hours after dosing on day 10
  Measured in nanomoles per liter (nmol/L).
tmax,0-24h,sema,Day10: Time to maximum semaglutide plasma concentration after the 10th dosing | From 0 to 24 hours after dosing on day 10
  Measured in hours (h).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com.
URL: http://novonordisk-trials.com